CLINICAL TRIAL: NCT05135936
Title: A Randomised Sham-controlled Study on the Effectiveness of Mild Water-filtered Infrared-A Whole-body Hyperthermia in Improving Symptoms and Quality of Life in Patients With Fibromyalgia Syndrome
Brief Title: Hyperthermia in Fibromyalgia Syndrome
Acronym: HYPAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jost Langhorst (Other)
Responsible Party: Sponsor-Investigator, Jost Langhorst, Prof., Universität Duisburg-Essen
Organization: Universität Duisburg-Essen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20079
Record Dates: First submitted 2021-04-13; First posted 2021-11-26 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Fibromyalgia
Keywords: hyperthermia; fibromyalgia syndrome; pain
MeSH Terms: conditions — Fibromyalgia; Hyperthermia; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Sham- and treatmentgroup
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperthermia Group (Experimental): For the study, the method of passive whole-body hyperthermia is used. The IRATHERM®1000 system (Von Ardenne Institute for Applied Medical Research/Dresden) is used, in which the entire body is heated to a core body temperature above the physiological 37°C. The aim is to achieve a core body temperature of 38.5°C within the framework of mild whole-body hyperthermia. After this warm-up phase, a temperature plateau phase of about 60 minutes follows, in which an attempt is made to maintain the core body temperature of 38.5°C. In the temperature plateau phase, a slight increase in the body core temperature is usually observed. The total time required for a session is given as 1.5 to 2 hours, but this depends on the individual constitution and daily condition of the patient and can be subject to fluctuations.
  Interventions: Behavioral: Hyperthermia Group
- Sham-Group (Sham Comparator): Within the patient information, privacy policy, etc., there is talk of "gentle hyperthermia" and classic, "mild hyperthermia". This serves to introduce the sham intervention as a control group compared to the patient. Lighting conditions, procedures, instructions and explanations are indistinguishable. Within the application, patients of the sham group will receive a hyperthermia application almost without overheating. In order to achieve this, the patients will be positioned on the IRATHERM®1000 in accordance with the Von Ardenne Institute's regulations. Due to the insulating blanket and the natural device and body heat, the patients of the sham group experience a gentle warmth, which is not the same as regular whole-body hyperthermia and an increase in the body core temperature of about 1.5 °C. In the sham setting, the core body temperature increases by about 0.3 to 0.4 °C within a 55-minute session.
  Interventions: Behavioral: Sham-Group

INTERVENTIONS:
Behavioral: Hyperthermia Group — The first hyperthermia treatment of the series is carried out for the second aptitude test, directly following the randomisation in the intervention group at the Hospital for Naturopathy and Integrative Medicine in Bamberg. The hyperthermia treatment is then carried out in a cycle of two treatments per week, with at least one day in between, over a period of three weeks, according to the manufacturer's instructions. According to the guidelines, the rectal (possibly vaginal) temperature (as body core temperature), heart rate and oxygen saturation (Sp02) are continuously determined during the hyperthermia treatment. During the treatment, continuous supervision by trained personnel is guaranteed, and a doctor is on call.
  Arms: Hyperthermia Group
Behavioral: Sham-Group — The number of treatments is equal to the number of treatments in the intervention group.
  Arms: Sham-Group

SUMMARY:
This study will examine the effectiveness of water-filtered whole-body hyperthermia during an outpatient setting in patients with fibromyalgia.

The duration of the study is about 3 weeks with two treatment units per week and a passive period (follow-up measurement) of 24 weeks after the outpatient setting.

DETAILED DESCRIPTION:
A total of about 40 participants over 18 years of age are sought, who will be divided into two groups of equal size after inclusion in the study. All participants will receive the same amount of water-filtered whole-body hyperthermia within the outpatient setting. One group receives the gentle form of GKHT, the other group receives the classic, mild GHKT. All abnormalities are documented by the responsible therapists, doctors and nurses. Changes in the area of pain and functional limitations as well as the intake of required medication are also recorded.

Before the start and after the completion of the studies, within the clinical stay, blood parameters were collected. In order to determine the secondary effectiveness of different questionnaire values are also collected. These are also documented after week 12 and after week 24, by means of telephone enquiries.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of fibromyalgia (FSQ)
* Pain VAS >= 4,0
* Signed declaration of consent

Exclusion Criteria:

* Participation in other clinical studies
* Contraindications for hyperthermia (severe cardiovascular diseases, tumour diseases, acute infections, pregnant and breastfeeding women)
* Acute and / or feverish microbial infections
* Patients with severe somatic, rheumatic concomitant endocrine or neurological diseases, in particular neurological diseases associated with cognitive disorders, severe liver or kidney and cardiac diseases
* Patients who are permanently treated with opioids, cannabis, immunosuppressive drugs (e.g. corticoids, immunosuppressants) or alpha/beta-A(nta)gonists due to a disease from the group described above
* Patients with pain due to a serious psychiatric illness (bipolar disorder, psychosis, personality disorder, severe depression, substance abuse) and serious systemic or neurological disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) - Intensity of pain (Numeric Rating Scale, NRS) | Week 0
  An inventory including 15 Items about the intensity of pain (4 items, numeric rating scales from 1 (no pain) to 10 (worst pain imaginable); primary outcome), pain impairment (7 items with NRS from 1-10) and the efficacy of medications/treatments.
Brief Pain Inventory (BPI) - Intensity of pain (Numeric Rating Scale, NRS) | Week 4
  An inventory including 15 Items about the intensity of pain (4 items, numeric rating scales from 1 (no pain) to 10 (worst pain imaginable); primary outcome), pain impairment (7 items with NRS from 1-10) and the efficacy of medications/treatments.

SECONDARY OUTCOMES:
Multidimensionl Fatigue Inventory (MFI-20) | Week 0
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue).
Multidimensionl Fatigue Inventory (MFI-20) | Week 4
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue).
Multidimensionl Fatigue Inventory (MFI-20) | Week 12
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue).
Multidimensionl Fatigue Inventory (MFI-20) | Week 30
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue).
Pittsburgh Sleep quality index (PSQI) | Week 0
  An inventory including 10 questions (plus subquestions) about the quality of sleep. Most of the questions range from ("Not during the past month" to "thee or more times a week"). The questions can be calculated in seven subscales.
Pittsburgh Sleep quality index (PSQI) | Week 4
  An inventory including 10 questions (plus subquestions) about the quality of sleep. Most of the questions range from ("Not during the past month" to "thee or more times a week"). The questions can be calculated in seven subscales.
Pittsburgh Sleep quality index (PSQI) | Week 12
  An inventory including 10 questions (plus subquestions) about the quality of sleep. Most of the questions range from ("Not during the past month" to "thee or more times a week"). The questions can be calculated in seven subscales.
Pittsburgh Sleep quality index (PSQI) | Week 30
  An inventory including 10 questions (plus subquestions) about the quality of sleep. Most of the questions range from ("Not during the past month" to "thee or more times a week"). The questions can be calculated in seven subscales.
Fibromyalgia Impact Questionnaire (FIQ) | Week 0
  An inventory measuring the disease-specific quality of life including 10 questions. The first question covers physical functioning ranging from 0 (always) to 3 (never). The second question is about wellbeing and the third examines the ability to work. Question 4-10 examine restrictions with visual analog scales (e.g. 0mm = not tired; 100mm = very tired) covering various symptoms like fatigue, anxiety or depression.
Fibromyalgia Impact Questionnaire (FIQ) | Week 4
  An inventory measuring the disease-specific quality of life including 10 questions. The first question covers physical functioning ranging from 0 (always) to 3 (never). The second question is about wellbeing and the third examines the ability to work. Question 4-10 examine restrictions with visual analog scales (e.g. 0mm = not tired; 100mm = very tired) covering various symptoms like fatigue, anxiety or depression.
Fibromyalgia Impact Questionnaire (FIQ) | Week 12
  An inventory measuring the disease-specific quality of life including 10 questions. The first question covers physical functioning ranging from 0 (always) to 3 (never). The second question is about wellbeing and the third examines the ability to work. Question 4-10 examine restrictions with visual analog scales (e.g. 0mm = not tired; 100mm = very tired) covering various symptoms like fatigue, anxiety or depression.
Fibromyalgia Impact Questionnaire (FIQ) | Week 30
  An inventory measuring the disease-specific quality of life including 10 questions. The first question covers physical functioning ranging from 0 (always) to 3 (never). The second question is about wellbeing and the third examines the ability to work. Question 4-10 examine restrictions with visual analog scales (e.g. 0mm = not tired; 100mm = very tired) covering various symptoms like fatigue, anxiety or depression.
Patient Global Impression of Change | Week 4
  One question about the patients global impression of change due to the therapy ranging from 1 (very much improved) to 7 (very much worse).
Patient Global Impression of Change | Week 12
  One question about the patients global impression of change due to the therapy ranging from 1 (very much improved) to 7 (very much worse).
Patient Global Impression of Change | Week 30
  One question about the patients global impression of change due to the therapy ranging from 1 (very much improved) to 7 (very much worse).
Pain Diary | Week -2-0
  Pain diary measuring the daily pain level at baseline. It also includes medication intakes, accompanying treatments and space for additional comments.
Pain Diary | Week 1-3
  Pain diary measuring the daily pain level during the period of intervention. It also includes medication intakes, accompanying treatments and space for additional comments.
Additional Treatments/Change of Medication | Week 12
  Record of additional treatments/change of medication to control for effects.
Additional Treatments/Change of Medication | Week 30
  Record of additional treatments/change of medication to control for effects.
Short-Form Mc Gill Pain Questionnaire - Deutsche Version (SF-MPQ-D) | Week 0
  The pain inventory includes three questions. The first one examines the quality of the pain with 15 items e.g. "throbbing", "shooting" raning from 0 (None) to 3 (severe). The second question examines the current level of pain with a visal analog scale (0mm= No Pain, 100mm= worst possible pain"). The third one examines the intensitiy of the whole pain experience (0=no Pain, 5 = excruciating).
Short-Form Mc Gill Pain Questionnaire - Deutsche Version (SF-MPQ-D) | Week 4
  The pain inventory includes three questions. The first one examines the quality of the pain with 15 items e.g. "throbbing", "shooting" raning from 0 (None) to 3 (severe). The second question examines the current level of pain with a visal analog scale (0mm= No Pain, 100mm= worst possible pain"). The third one examines the intensitiy of the whole pain experinece (0=no Pain, 5 = excruciating).
Short-Form Mc Gill Pain Questionnaire - Deutsche Version (SF-MPQ-D) | Week 12
  The pain inventory includes three questions. The first one examines the quality of the pain with 15 items e.g. "throbbing", "shooting" raning from 0 (None) to 3 (severe). The second question examines the current level of pain with a visal analog scale (0mm= No Pain, 100mm= worst possible pain"). The third one examines the intensitiy of the whole pain experience (0=no Pain, 5 = excruciating).
Short-Form Mc Gill Pain Questionnaire - Deutsche Version (SF-MPQ-D) | Week 30
  The pain inventory includes three questions. The first one examines the quality of the pain with 15 items e.g. "throbbing", "shooting" raning from 0 (None) to 3 (severe). The second question examines the current level of pain with a visal analog scale (0mm= No Pain, 100mm= worst possible pain"). The third one examines the intensitiy of the whole pain experience (0=no Pain, 5 = excruciating).
age | Week 0
  age in years
sex | Week 0
  identification of gender
height | Week 0
  in meters
weight | Week 0
  in kg
marital status | Week 0
  identification of marital status
education | Week 0
  identification of the educational level
job | Week 0
  identification of the current job (4 questions about job/application for pension)
G-EEE (Generic Rating for Treatment pre-experiences, Treatment Expectations and Treatment effects) | Week 0
  A non validated inventory including 11 items measuring pre-experiences, treatment expectations and treatment effects.
G-EEE (Generic Rating for Treatment pre-experiences, Treatment Expectations and Treatment effects) | Week 4
  A non validated inventory including 11 items measuring pre-experiences, treatment expectations and treatment effects.
G-EEE (Generic Rating for Treatment pre-experiences, Treatment Expectations and Treatment effects) | Week 12
  A non validated inventory including 11 items measuring pre-experiences, treatment expectations and treatment effects.
G-EEE (Generic Rating for Treatment pre-experiences, Treatment Expectations and Treatment effects) | Week 30
  A non validated inventory including 11 items measuring pre-experiences, treatment expectations and treatment effects.
SF-36 health survey | Week 0
  An inventory including 36 item measuring the current health status and generic quality of life of the patients. It includes eight subscales, that can be summarized in one physical and one psychological summary scale.
SF-36 health survey | Week 4
  An inventory including 36 item measuring the current health status and generic quality of life of the patients. It includes eight subscales, that can be summarized in one physical and one psychological summary scale.
SF-36 health survey | Week 12
  An inventory including 36 item measuring the current health status and generic quality of life of the patients. It includes eight subscales, that can be summarized in one physical and one psychological summary scale.
SF-36 health survey | Week 30
  An inventory including 36 item measuring the current health status and generic quality of life of the patients. It includes eight subscales, that can be summarized in one physical and one psychological summary scale.
Shortform of PHQ-D (Patient Health Questionnaire) | Week 0
  An inventory measurung the psychological health status including among others 9 items about depression (PHQ-9), 15 items about somatization (PHQ-15) and 7 items about general anxietey (GAD-7).
Shortform of PHQ-D (Patient Health Questionnaire) | Week 4
  An inventory measurung the psychological health status including among others 9 items about depression (PHQ-9), 15 items about somatization (PHQ-15) and 7 items about general anxietey (GAD-7).
Shortform of PHQ-D (Patient Health Questionnaire) | Week 12
  An inventory measurung the psychological health status including among others 9 items about depression (PHQ-9), 15 items about somatization (PHQ-15) and 7 items about general anxietey (GAD-7).
Shortform of PHQ-D (Patient Health Questionnaire) | Week 30
  An inventory measurung the psychological health status including among others 9 items about depression (PHQ-9), 15 items about somatization (PHQ-15) and 7 items about general anxietey (GAD-7).
Brief Pain Inventory (BPI) - Intensity of pain (Numeric Rating Scale, NRS) | Week 12
  An inventory including 15 Items about the intensity of pain (4 items, numeric rating scales from 1 (no pain) to 10 (worst pain imaginable), pain impairment (7 items with NRS from 1-10) and the efficacy of medications/treatments.
Brief Pain Inventory (BPI) - Intensity of pain (Numeric Rating Scale, NRS) | Week 30
  An inventory including 15 Items about the intensity of pain (4 items, numeric rating scales from 1 (no pain) to 10 (worst pain imaginable), pain impairment (7 items with NRS from 1-10) and the efficacy of medications/treatments.
Patient Interview | Week 12
  Qualitative telephone interviews with 10 patients of the mild whole body hyperthermia group (Experimental group) to get detailed experiences of the patients (30-45 min).
Adverse events (AE) | Week 1-3
  Description of adverse events during the interventions by therapists.

OTHER OUTCOMES:
Blood count | Week 0
  (to measure baseline status)
Blood count | Week 3 - after last intervention
  (to measure acute effects)
Blood count | Week 4
  (to measure acute effects)
C-reactive Protein (CRP) | Week 0
  Level of c-reactive protein (CRP) in blood to measure inflammation.
C-reactive Protein (CRP) | Week 3 - after last intervention
  Level of c-reactive protein (CRP) in blood to measure inflammation (to measure acute effects).
C-reactive Protein (CRP) | Week 4
  Level of c-reactive protein (CRP) in blood to measure inflammation.
Blood cell sedimenation rate (BSG) | Week 0
  Serum parameter.
Blood cell sedimenation rate (BSG) | Week 3 - after last intervention
  Serum parameter (to measure acute effects).
Blood cell sedimenation rate (BSG) | Week 4
  Serum parameter.
Coagulation | Week 0
  Coagulation measured in blood.
Coagulation | Week 3 - after last intervention
  Coagulation measured in blood.
Coagulation | Week 4
  Coagulation measured in blood.
Tumor Necrosis Factor (TNF-α) | Week 0
  Serum parameter.
Tumor Necrosis Factor (TNF-α) | Week 3 - after last intervention
  Serum parameter.
Tumor Necrosis Factor (TNF-α) | Week 4
  Serum parameter.
Interleukin-1 (IL-1) | Week 0
  Serum parameter (Zytokines).
Interleukin-1 (IL-1) | Week 3 - after last intervention
  Serum parameter (Zytokines).
Interleukin-1 (IL-1) | Week 4
  Serum parameter (Zytokines).
Interleukin-6 (IL-6) | Week 0
  Serum parameter (Zytokines).
Interleukin-6 (IL-6) | Week 3 - after last intervention
  Serum parameter (Zytokines).
Interleukin-6 (IL-6) | Week 4
  Serum parameter (Zytokines).
Interleukin-8 (IL-8) | Week 0
  Serum parameter (Zytokines).
Interleukin-8 (IL-8) | Week 3 - after last intervention
  Serum parameter (Zytokines).
Interleukin-8 (IL-8) | Week 4
  Serum parameter (Zytokines).
Interleukin-10 (IL-10) | Week 0
  Serum parameter (Zytokines).
Interleukin-10 (IL-10) | Week 3 - after last intervention
  Serum parameter (Zytokines).
Interleukin-10 (IL-10) | Week 4
  Serum parameter (Zytokines).
creatinine | Week 4
  Serum parameter.
GOT, GPT, GGT | Week 4
  Serum Parameters - Liver enzymes.

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, Prof., Study Director — Sozialstiftung Bamberg
Locations (1):
- Sozialstiftung Bamberg, Klinik für Intergrative Medizin, Bamberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No